CLINICAL TRIAL: NCT03824860
Title: Yoga for Painful Chemotherapy-Induced Peripheral Neuropathy: A Pilot, Randomized-Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Robert Knoerl, PhD, RN, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-578
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Yoga; Chronic Pain; Neuropathic Pain
Keywords: Chemotherapy-induced Peripheral Neuropathy; Yoga; Chronic Pain; Neuropathic Pain
MeSH Terms: conditions — Chronic Pain; Neuralgia | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Program (Experimental): Eight-weeks, therapist and self-guided yoga
  Interventions: Behavioral: Yoga
- Treatment as usual (No Intervention): Control group participants will continue to receive usual care and symptom management strategies from clinicians during the study.

INTERVENTIONS:
Behavioral: Yoga — Participants will attend at least one group class per week (in-person or Zoom) and practice one self-guided yoga video class at home on their own per week, over eight weeks
  Participants may choose to attend "Flow Yoga" and/or "Chair Flow Yoga" classes. These classes will be videotaped and made available to participants electronically.
  Classes consist of:
  * guided breathing exercises,
  * upper and lower extremity stretching
  * structured postures and movements to improve balance and strength
  Arms: Yoga Program

SUMMARY:
This research study will examine the feasibility of conducting an eight-week yoga intervention for individuals with chronic painful chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
This research study will examine the feasibility of conducting an eight-week yoga intervention for individuals with chronic painful chemotherapy-induced peripheral neuropathy. The investigators will also explore participants' perceptions of acceptability and satisfaction with the yoga intervention. Lastly, the investigators will examine changes in chemotherapy-induced peripheral neuropathy severity, physical function, sleep-related impairment, fatigue, anxiety, depression, and pain following the eight-week yoga intervention.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age,

* self-report ≥ 4/10 worst chemotherapy-induced peripheral neuropathy pain over the past week,
* at least three months post neurotoxic chemotherapy completion
* signed informed consent,
* willingness to participate in all study activities
* speak/read English

Exclusion Criteria:

* prognosis of less than three months,
* documented peripheral neuropathy due to other causes (e.g., diabetes),
* planned receipt of neurotoxic chemotherapy during the study period,
* practice yoga >45 minutes per week over the past six months,
* diagnosis or documented recent history of significant psychiatric comorbidity (i.e., psychosis, suicidal ideation, or substance abuse)
* clinician deems that the patient is physically/functionally unable to participate in a yoga program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited to participate in the study | From enrollment to end of treatment at 8 weeks.
  Feasibility of participant recruitment to the study
Frequency of yoga practice by participants | From enrollment to end of treatment at 8 weeks.
  Feasibility of participant adherence to the yoga intervention
Frequency of outcome assessments completed by participants. | From enrollment to end of treatment at 8 weeks.
  Feasibility of participant adherence to outcome assessments

SECONDARY OUTCOMES:
Acceptability and Satisfaction with Participation in Yoga Intervention | At the end of treatment, 8 weeks after enrollment
  We will use semi-structured interviews to gain information about participants' experience with the yoga program
Worst Chemotherapy-Induced Peripheral Neuropathy Pain Intensity | At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in 0 - 10 numerical rating scale of worst chemotherapy-induced peripheral neuropathy pain (via 7-day pain diary) from enrollment to end of treatment at 8 weeks. Total scores range from 0 - 10, with higher scores representing worse pain.
Chemotherapy-Induced Peripheral Neuropathy Severity | From enrollment to end of treatment at 8 weeks.At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in European Organization of Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy Scale-20 score from enrollment to end of treatment at 8 weeks. Total scores range from 0 - 100, with higher scores representing worse chemotherapy-induced peripheral neuropathy severity.
Pain Interference | At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4a score from enrollment to the end of treatment at 8 weeks. Total scores range from 41.6 - 75.6, with higher scores representing worse pain interference.
Sleep-Related Impairment | At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Sleep-related Impairment 8a score from enrollment to the end of treatment at 8 weeks. Total scores range from 30.0 - 80.1 with higher scores representing worse sleep-related impairment.
Anxiety assessed by the "Change in Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety" | At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety 4a score from enrollment to the end of treatment at 8 weeks. Total scores range from 40.3 - 81.6, with higher scores representing worse anxiety.
Depression assessed by Change in Patient Reported Outcomes Measurement Information System (PROMIS) Depression | At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Depression 4a score from enrollment to the end of treatment at 8 weeks. Total scores range from 41.0 - 79.4, with higher scores representing worse depression.
Fatigue assessed by Change in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue | At the time of enrollment and at the end of treatment, 8 weeks after enrollment
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue 4a score from enrollment to the end of treatment at 8 weeks. Total scores range from 33.7 - 75.8, with higher scores representing worse fatigue.
Physical Function | At the time of enrollment and at the end of treatment, at 8 weeks.
  Change in Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function 4a score from enrollment to the end of treatment at 8 weeks. Total scores range from 22.5 - 57.0, with higher scores representing better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Robert Knoerl, PhD; Study PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Brigham and Women's Hospital - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Knoerl R, Giobbie-Hurder A, Berfield J, Berry D, Meyerhardt JA, Wright AA, Ligibel JA. Yoga for chronic chemotherapy-induced peripheral neuropathy pain: a pilot, randomized controlled trial. J Cancer Surviv. 2022 Aug;16(4):882-891. doi: 10.1007/s11764-021-01081-z. Epub 2021 Sep 15. PMID 34524631
- [Derived] Knoerl R, Phillips CS, Berfield J, Woods H, Acosta M, Tanasijevic A, Ligibel J. Lessons learned from the delivery of virtual integrative oncology interventions in clinical practice and research during the COVID-19 pandemic. Support Care Cancer. 2021 Aug;29(8):4191-4194. doi: 10.1007/s00520-021-06174-0. Epub 2021 Mar 26. PMID 33772364

DOCUMENTS (1):
  • Informed Consent Form (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03824860/ICF_000.pdf